CLINICAL TRIAL: NCT05670041
Title: Re-hospitalisation After Transcatheter Aortic Valve Implantation
Acronym: HOSPITAVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ole De Backer (Other)
Responsible Party: Sponsor-Investigator, Ole De Backer, Professor, dr. med., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H-21036155
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Aortic Valve Disease; Aortic Valve Stenosis
Keywords: Transcatheter Aortic Valve Implantation; Transcatheter Aortic Valve Replacement; Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard follow-up (No Intervention)
- Intensified follow-up (Experimental): Early, intensified follow-up after discharge from TAVI-procedure consisting of telephone consults and an additional visit to the outpaitent clinic.
  Interventions: Behavioral: Intensified follow-up

INTERVENTIONS:
Behavioral: Intensified follow-up — Early, intensified follow-up after discharge from TAVI-procedure.
  Arms: Intensified follow-up

SUMMARY:
The goal of this study is to investigate whether patient-tailored follow-up for patients treated with transcatheter aortic valve implantation (TAVI) can prevent re-hospitalisation and improve quality of life compared with the standard follow-up program.

The rationale of this study is the persistently high rate of re-hospitalisation after TAVI, which increases the risk of mortality and diminishes the patient-evaluated quality of life. Our hypothesis is that patient-tailored follow-up for patients treated with TAVI will reduce the rate of re-hospitalisation after the TAVI-procedure and improve quality of life.

The primary endpoints are the rate of re-hospitalisation within 90 days of the procedure and quality of life adjusted life years at 90-day follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent technical successful TAVI
* Residing in Denmark
* Provided written informed consent

Exclusion Criteria:

* Index admission mortality
* Index admission conversion to open surgery
* Age < 18 years
* Women of childbearing potential, pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2024-03-16 (Estimated); Study Completion 2025-03-16 (Estimated)

PRIMARY OUTCOMES:
The rate of all-cause hospitalisations between discharge from the index procedure and 90 days post-TAVI | 365 days
  Primary safety endpoint
Quality-of-life adjusted life years at 90 days after the TAVI-procedure | 365 days
  Primary efficacy endpoint

SECONDARY OUTCOMES:
The risk of all-cause mortality | 365 days

CONTACTS AND LOCATIONS:
Overall Officials: Lars Sondergaard, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Baekke PS, Jorgensen TH, Bieliauskas G, Sondergaard L, De Backer O. Impact of Intensified Outpatient Follow-Up on Rehospitalization After Transcatheter Aortic Valve Implantation: Results From the HOSPITAVI Trial. Am J Cardiol. 2025 Jun 15;245:17-24. doi: 10.1016/j.amjcard.2025.01.031. Epub 2025 Feb 1. PMID 39900323